CLINICAL TRIAL: NCT05214976
Title: A Phase Ⅰb/Ⅱ Clinical Study on the Open-label and Multiple Centers of Camrelizumab for Injection in Combination With Famitinib Malate Capsule and Paclitaxel For Injection(Albumin Bound) in Advanced Solid Tumors of Patients
Brief Title: A Trial of Camrelizumab for Injection in Combination With Famitinib Malate Capsule and Paclitaxel For Injection(Albumin Bound) in Advanced Solid Tumors of Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-II-222
Record Dates: First submitted 2022-01-28; First posted 2022-01-31 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — camrelizumab; Injections; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Camrelizumab for Injection in combination with Famitinib malate capsule and Paclitaxel
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Experimental)
  Interventions: Drug: Camrelizumab for Injection, Famitinib malate capsule, Paclitaxel For Injection(Albumin Bound)

INTERVENTIONS:
Drug: Camrelizumab for Injection, Famitinib malate capsule, Paclitaxel For Injection(Albumin Bound) — Firstly Dose Escalation of Camrelizumab for Injection in combination with Famitinib malate capsule and Paclitaxel For Injection(Albumin Bound) should be conducted. According to the DLT data in the dose escalation period, dosage of Famitinib malate capsule or Paclitaxel For Injection(Albumin Bound) would be adjusted. After dose escalation period, in order to evaluate the tolerance, study would choose the dosage regimen to complete the Dose Expansion period. The indication expansion would be conducted after that. The study would select specific indications based on the previous efficacy data with the RP2D of the combination therapy.

SUMMARY:
The study is being conducted to evaluate safety, tolerability and preliminary efficacy of Camrelizumab for Injection in combination with Famitinib malate capsule and Paclitaxel For Injection(Albumin Bound) for advanced solid tumors of patients. To explore the reasonable dosage of dosage regimen of combination therapy for advanced malignant tumors of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years and ≤75 years at the time of signing the ICF;
2. Dose Escalation Period: Histopathologically documented incurable advanced malignancies with standard treatment failure;
3. At least one measurable lesion that meets RECIST 1.1 criteria in case of solid tumors;
4. An Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1;
5. Life expectancy ≥3 months;
6. Adequate organ functions as defined;
7. Ability to understand and voluntarily agrees to participate by giving written informed consent for the study.

Exclusion Criteria:

1. The imaging examinations shows the tumor invades large blood vessels; Or as the assessment of the investigator, the tumor is highly likely to invade important blood vessels which would cause fatal bleeding during treatment;
2. The imaging examinations shows significant pulmonary cavitary tumors occurs with the bleeding risk as the investigator's assessment;
3. patients with active brain metastasis (without medical control or with clinical symptoms), cancerous meningitis, or spinal cord compression;
4. Uncontrollable pleural effusion, pericardial effusion or peritoneal effusion, with clinical symptoms;
5. Severe bong injury caused by metastatic tumor of bone;
6. Prior malignancy (other than current malignant tumor) within 3 years before the first dose of study treatment;
7. History of autoimmune diseases;
8. Evidence or history of arterial/venous thrombosis within 6 months before the first dose;
9. Patients with interstitial pneumonitis or interstitial lung disease; past history of interstitial pneumonitis or interstitial lung disease requiring hormone therapy;
10. When receiving immune checkpoint inhibitors previously, myocarditis related with immune, ≥ grade 2 of pneumonia related with immune or ≥ grade 3 of other adverse reactions related with immune occurred.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity | first dose of study medication up to 21 days]
  Dose Limited Toxicity of Camrelizumab for Injection in combination with Famitinib malate capsule and Paclitaxel For Injection(Albumin Bound)
Recommended phase II dose | first dose of study medication up to 21 days
  The Recommended phase II dose of Camrelizumab for Injection in combination with Famitinib malate capsule and Paclitaxel For Injection(Albumin Bound)
ORR | from the date of the first dose to the date of disease progression evaluated based on RECIST v1.1 criteria, or initiation of other anti-tumor treatment, whichever occurs first, up to 6 months
  Objective Response Rate, Efficacy endpoints of Camrelizumab for Injection in combination with Famitinib malate capsule and Paclitaxel For Injection(Albumin Bound) in Advanced Solid Tumors of Patients

SECONDARY OUTCOMES:
DoR | from the date of the firstly documented tumor response (evaluated based on RECIST v1.1 criteria) to the date of the firstly documented disease progression (evaluated based on RECIST v1.1 criteria) or the date of death for any reason, up to 6 months
  Duration of response, Efficacy endpoints of Camrelizumab for Injection in combination with Famitinib malate capsule and Paclitaxel For Injection(Albumin Bound) in Advanced Solid Tumors of Patients
DCR | from the date of the first dose to the date of the firstly documented disease progression (evaluated based on RECIST v1.1 criteria) or the date of death for any reason, up to 6 months
  Disease control rate, Efficacy endpoints of Camrelizumab for Injection in combination with Famitinib malate capsule and Paclitaxel For Injection(Albumin Bound) in Advanced Solid Tumors of Patients
PFS | from the date of the first dose to the date of the firstly documented disease progression (evaluated based on RECIST v1.1 criteria) or the date of death for any reason, up to 6 months
  Progression-free survival, Efficacy endpoints of Camrelizumab for Injection in combination with Famitinib malate capsule and Paclitaxel For Injection(Albumin Bound) in Advanced Solid Tumors of Patients
OS | from the date of the first dose to the date of death for any reason, up to 100 months
  Overall survival, Efficacy endpoints of Camrelizumab for Injection in combination with Famitinib malate capsule and Paclitaxel For Injection(Albumin Bound) in Advanced Solid Tumors of Patients
12 months' survival rate | from the date of the first dose up to 12 months
  Efficacy endpoints of Camrelizumab for Injection in combination with Famitinib malate capsule and Paclitaxel For Injection(Albumin Bound) in Advanced Solid Tumors of Patients
TTF | from the date of the first dose to the date of treatment termination, up to 6 months
  Time to Failure, Efficacy endpoints of Camrelizumab for Injection in combination with Famitinib malate capsule and Paclitaxel For Injection(Albumin Bound) in Advanced Solid Tumors of Patients
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) | from signature completion of ICF to 90 days after the last dose or to the beginning of the new anti-cancer therapy, up to 6 months
  Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
The occurrence rate of dose titration | from signature completion of ICF to 90 days after the last dose or to the beginning of the new anti-cancer therapy, up to 6 months
  The occurrence rate of dose interruption, dose decrease and dose termination because of study drug related toxicity during the study
concentration of drug in serum | 0.5 hour before first dose of Camrelizumab for Injection to 30 days after last dose
  PK concentration of Camrelizumab for Injection
concentration of drug in plasma | 2 days before first dose of Camrelizumab for Injection to 1 hour before the first dose of tenth cycle of Famitinib malate capsule
  PK concentration of Famitinib malate capsule and its intermediate metabolite, and Paclitaxel For Injection(Albumin Bound)
Tmax | 2 days before first dose of Camrelizumab for Injection to 1 hour before the first dose of tenth cycle of Famitinib malate capsule
  PK parameters of Famitinib malate capsule and its intermediate metabolite, and Paclitaxel For Injection(Albumin Bound)
Cmax | 2 days before first dose of Camrelizumab for Injection to 1 hour before the first dose of tenth cycle of Famitinib malate capsule
  PK parameters of Famitinib malate capsule and its intermediate metabolite, and Paclitaxel For Injection(Albumin Bound)
AUC | 2 days before first dose of Camrelizumab for Injection to 1 hour before the first dose of tenth cycle of Famitinib malate capsule
  PK parameters of Famitinib malate capsule and its intermediate metabolite, and Paclitaxel For Injection(Albumin Bound)
t1/2 | 2 days before first dose of Camrelizumab for Injection to 1 hour before the first dose of tenth cycle of Famitinib malate capsule
  PK parameters of Famitinib malate capsule and its intermediate metabolite, and Paclitaxel For Injection(Albumin Bound)
CL/F | 2 days before first dose of Camrelizumab for Injection to 1 hour before the first dose of tenth cycle of Famitinib malate capsule
  PK parameters of Famitinib malate capsule and its intermediate metabolite, and Paclitaxel For Injection(Albumin Bound)
ADA | the date of first dose up to 30 days after last dose
  Anti-drug antibody, Immunogenicity of Camrelizumab for Injection
NAb | the date of first dose up to 30 days after last dose
  Neutralizing Antibody, Immunogenicity of Camrelizumab for Injection

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided